CLINICAL TRIAL: NCT03055403
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Continuous Intravenous Injection, Dose Escalation, Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of M201-A in Healthy Japanese Subjects
Brief Title: First-in-Human Dose Escalation Study of M201-A in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuji KUMAGAI (Other)
Collaborators: Aetas Pharma Co. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yuji KUMAGAI, Professor, Kitasato University
Organization: Kitasato University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M201-A-CT-001
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M201-A Injection (Experimental): Active Substance: M201-A Route of administration: continuous intravenous injection
  Interventions: Drug: M201-A Injection
- Placebo (Placebo Comparator): Saline Placebo for M201-A Route of administration: continuous intravenous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M201-A Injection — Active Substance: M201-A Route of administration: continuous intravenous injection
  Arms: M201-A Injection
Drug: Placebo — Saline Placebo for M201-A Route of administration: continuous intravenous injection
  Arms: Placebo

SUMMARY:
This Phase I first-in-human is designed to evaluate the safety, tolerability and pharmacokinetics of single ascending doses of M201-A administered by single continuous intravenous injection in Healthy Japanese subjects.

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

* Japanese Healthy Male subjects
* Age 20 to less than 40 years of age
* Body Mass Index (BMI) of 18.5 to less than 25.0 kg/m2
* Written informed consent must be obtained on a voluntary basis before any assessment is performed.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

* Presence or past medical history of hepatic impairments, renal impairments, cardiovascular disease, gastrointestinal disease and others which are inappropriate for participating in this clinical trial
* Past medical history of cancer, cerebral infarction or cardiac infarction
* Presence or past medical history of allergic reactions or idiosyncrasies to food, medicinal substance and metallic materials
* QTcF > 450ms at the screening examination
* NT-proBNP > 125 pg/mL at the screening examination
* Any risk factors of Torsades de Pointes including such as heart failure, hypokalemia, long QT interval syndrome due to family medical history

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Throughout the study duration (up to day8)
  adverse events, serious adverse events, physical examinations, vital sign measurements, 12-lead ECGs, Holter ECG, clinical laboratory safety tests (including hematology, chemistry, and urinalysis), recording of concomitant medications and procedures.

SECONDARY OUTCOMES:
Pharmacokinetics-Cmax | Predose, 0, 5, 15, 30, 60, 120, 240, 480 minutes and 24 hours after the IV infusion of M201-A
  Observed maximum plasma concentration (Cmax) of M201-A
Pharmacokinetics-Tmax | Predose, 0, 5, 15, 30, 60, 120, 240, 480 minutes and 24 hours after the IV infusion of M201-A
  Time to Cmax (Tmax) of M201-A
Pharmacokinetics-AUC0-24 | Predose, 0, 5, 15, 30, 60, 120, 240, 480 minutes and 24 hours after the IV infusion of M201-A
  Area under the plasma concentration-time curve from time zero to 24hour of M201-A
Pharmacokinetics-AUC0-t | Predose, 0, 5, 15, 30, 60, 120, 240, 480 minutes and 24 hours after the IV infusion of M201-A
  -Area under the plasma concentration-time curve calculated from time zero to the last measured time point (AUC0-t) of M201-A
Pharmacokinetics-AUC0-∞ | Predose, 0, 5, 15, 30, 60, 120, 240, 480 minutes and 24 hours after the IV infusion of M201-A
  Area under the plasma concentration-time curve calculated from time zero to infinity (AUC0-∞) of M201-A
Pharmacokinetics-t1/2 | Predose, 0, 5, 15, 30, 60, 120, 240, 480 minutes and 24 hours after the IV infusion of M201-A
  Elimination half-life (t1/2) of M201-A
Pharmacokinetics-CL | Predose, 0, 5, 15, 30, 60, 120, 240, 480 minutes and 24 hours after the IV infusion of M201-A
  Apparent clearance of drug from plasma (CL) of M201-A
Pharmacokinetics-Vd | Predose, 0, 5, 15, 30, 60, 120, 240, 480 minutes and 24 hours after the IV infusion of M201-A
  Apparent volume of distribution during the terminal phase (Vd) of M201-A
Pharmacokinetics-E0-24 | up to 24 hours
  Amount of drug excreted in urine from time zero to 24hour of M201-A
Pharmacokinetics-Ae | up to 24 hours
  Urinary excretion rate of M201-A

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Kitasato University Hospital, THE KITASATO INSTITUTE, Sagamihara, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No